CLINICAL TRIAL: NCT01677871
Title: Study of Efficacy and Safety of Modified Anti-tubercular Regimens in Treatment of Tuberculosis in Patients With Underlying Compensated and Decompensated Chronic Liver Disease
Brief Title: Efficacy and Safety of Modified Anti-tubercular Regimens in Treatment of Tuberculosis in Patients With Underlying Compensated and Decompensated Chronic Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ATT-01
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Liver Disease With Tuberclosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2HRZE/4HR (Experimental): Isoniazid + Rifampicin+Pyrazinamide+Ethambutol for initial 2 months floolowed by Isoniazid + Rifampicin for next 4 months
  Interventions: Drug: 2HRLE/4HR
- 2HRLE/4HR (Active Comparator): Isoniazid + Rifampicin+ Levofloxacin+Ethambutol for initial 2 months followed by Isonizid + Rifampicin for next 4 months
  Interventions: Drug: 2HRZE/4HR
- 9HLE (Experimental): Isoniazid+ Levofloxacin+ Ethambutol for 9 months
  Interventions: Drug: 9RLE
- 9RLE (Active Comparator): Rifampicin + Levofloxacin+ Ethambutol for 9 months
  Interventions: Drug: 9HLE

INTERVENTIONS:
Drug: 2HRZE/4HR — Isoniazid + Rifampicin+Pyrazinamide+Ethambutol for initial 2 months floolowed by Isoniazid + Rifampicin for next 4 months
  Arms: 2HRLE/4HR
Drug: 2HRLE/4HR — Isoniazid + Rifampicin+ Levofloxacin+Ethambutol for initial 2 months followed by Isonizid + Rifampicin for next 4 months
  Arms: 2HRZE/4HR
Drug: 9HLE — Isoniazid+ Levofloxacin+ Ethambutol for 9 months
  Arms: 9RLE
Drug: 9RLE — Rifampicin + Levofloxacin+ Ethambutol for 9 months
  Arms: 9HLE

SUMMARY:
During the Study:

* Subject is required to visit every week for the first 2 months and then every month till completion of study or as and when required
* The usual symptomatic and supportive treatment of Chronic Liver Disease, including use of antiviral, will be given to all patients.
* Effort will be made to avoid use of other hepatotoxic drug(s) during Anti-Tubercular Treatment.
* Liver function tests (LFT) will be done weekly during first 2 months then at one month interval or as when required.
* The treatment efficacy of Anti-Tubercular Treatment (ATT) will be made on the basis of clinical, biochemical, microbiological and imaging parameters at months 2, 4, 7 and 9. Patients not improving at 4 weeks after initiation of treatment will be shifted to alternative regimens and will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females subjects aged 18-75 years.
* Subjects with chronic liver disease (cirrhosis)
* Pulmonary or extra-pulmonary tuberculosis.
* Serum ALT≤5times upper limit and serum bilirubin ≤3 mg/dl.
* consent and willingness to follow-up

Exclusion Criteria:

* Serum ALT>5times upper limit and serum bilirubin >3 mg/dl.
* Renal failure (serum creatinine>2mg/dl).
* Presence of hepatocellular carcinoma
* Alcoholic cirrhotic who continue to drink alcohol.
* Prior history of ATT (ANTI TUBERCULAR TREATMENT) with documented hepatotoxicity.
* Known hypersensitivity to levofloxacin, other quinolones

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Successful completion of modified ATT (ANTI TUBERCULAR TREATMENT) regimen. | 6 and 9 months

SECONDARY OUTCOMES:
Worsening of CTP (CHILD TURCOTTE PUGH) score to ≥10 for patients with compensated cirrhosis, | 6 and 9 months
Failure to re-institute the assigned ATT (ANTI TUBERCULAR TREATMENT) regimen after development of an episode of hepatotoxicity. (I.e. second episode of hepatotoxicity.
Survival | 6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Naveen Kumar, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India